CLINICAL TRIAL: NCT00054860
Title: A Phase I Dose-Escalation Clinical Trial to Evaluate the Safety and Immunogenicity of the EP HIV-1090 DNA Vaccine in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Safety of and Immune System Response to an HIV Vaccine (EP HIV-1090) in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 048; 10197 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2003-02-11; First posted 2003-02-13 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; HIV Seronegativity; HIV-1; AIDS Vaccines; Vaccines, DNA; Dose-Response Relationship, Immunologic; CD4-Positive T-Lymphocytes; CD8-Positive T-Lymphocytes; Epitopes
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: EP HIV-1090

SUMMARY:
The purpose of this study is to test the safety of an HIV DNA vaccine (EP HIV-1090) and to test whether or not the vaccine can stimulate immune system responses in HIV uninfected people. This vaccine uses only parts of the virus's DNA and cannot cause HIV infection.

DETAILED DESCRIPTION:
Epidemiological and animal model data support the hypothesis that HIV specific cytotoxic T lymphocyte (CTL) responses contribute to control and clearance of the virus. Vaccines designed specifically to induce CTL responses are likely to be well suited for protection against HIV infection and disease progression. EP HIV-1090 is a DNA vaccine composed of 21 highly specific CTL epitopes. The vaccine is designed to optimize the immune response in people expressing one of three HLA Class I antigen subtypes: HLA-A2, -A3, and -B7. This design is predicted to induce an immune response in 85% of individuals in the general population. There is also a helper T lymphocyte (HTL) facilitating epitope (PADRE) in the vaccine. The vaccine is formulated with a water soluble polymer (polyvinylpyrrolidone) that protects the DNA and facilitates cellular uptake. This study will assess the safety of and immune response to different doses of EP HIV-1090 in healthy, HIV uninfected adults.

Participants in this study will be randomized to receive either one of three different doses of vaccine or placebo. Participants will receive vaccinations or placebo at study entry and Months 1, 3, and 6. Both vaccinations and placebo are administered by intramuscular injection. Participants will be followed for 18 months and will have 12 study visits. Each study visit will include a physical exam, medical history, and blood and urine tests. Each participant will have four HIV tests during the study. Women will have at least five pregnancy tests during the study.

ELIGIBILITY:
Inclusion Criteria

* HIV negative
* Positive for one or more of the following HLA supertypes: -A2, -A3, or -B7
* Willing to receive HIV test results
* Good general health
* Acceptable methods of contraception for females of reproductive potential
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV is positive

Exclusion Criteria

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Active syphilis
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Unstable asthma
* Type 1 or Type 2 Diabetes Mellitus
* Thyroid disease requiring treatment
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey J. Gorse, MD, Study Chair — St. Louis University
Locations (5):
- United States (4):
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - Miriam Hospital's HVTU, Providence, Rhode Island
- Gaborone Prevention/Treatment Trials CRS, Gaborone, Botswana

REFERENCES:
- [Background] Sette A, Vitiello A, Reherman B, Fowler P, Nayersina R, Kast WM, Melief CJ, Oseroff C, Yuan L, Ruppert J, Sidney J, del Guercio MF, Southwood S, Kubo RT, Chesnut RW, Grey HM, Chisari FV. The relationship between class I binding affinity and immunogenicity of potential cytotoxic T cell epitopes. J Immunol. 1994 Dec 15;153(12):5586-92. PMID 7527444
- [Background] Altfeld MA, Livingston B, Reshamwala N, Nguyen PT, Addo MM, Shea A, Newman M, Fikes J, Sidney J, Wentworth P, Chesnut R, Eldridge RL, Rosenberg ES, Robbins GK, Brander C, Sax PE, Boswell S, Flynn T, Buchbinder S, Goulder PJ, Walker BD, Sette A, Kalams SA. Identification of novel HLA-A2-restricted human immunodeficiency virus type 1-specific cytotoxic T-lymphocyte epitopes predicted by the HLA-A2 supertype peptide-binding motif. J Virol. 2001 Feb;75(3):1301-11. doi: 10.1128/JVI.75.3.1301-1311.2001. PMID 11152503
- [Background] Woodberry T, Gardner J, Mateo L, Eisen D, Medveczky J, Ramshaw IA, Thomson SA, Ffrench RA, Elliott SL, Firat H, Lemonnier FA, Suhrbier A. Immunogenicity of a human immunodeficiency virus (HIV) polytope vaccine containing multiple HLA A2 HIV CD8(+) cytotoxic T-cell epitopes. J Virol. 1999 Jul;73(7):5320-5. doi: 10.1128/JVI.73.7.5320-5325.1999. PMID 10364278
- [Background] Livingston BD, Newman M, Crimi C, McKinney D, Chesnut R, Sette A. Optimization of epitope processing enhances immunogenicity of multiepitope DNA vaccines. Vaccine. 2001 Sep 14;19(32):4652-60. doi: 10.1016/s0264-410x(01)00233-x. PMID 11535313
- [Background] Hanke T, Samuel RV, Blanchard TJ, Neumann VC, Allen TM, Boyson JE, Sharpe SA, Cook N, Smith GL, Watkins DI, Cranage MP, McMichael AJ. Effective induction of simian immunodeficiency virus-specific cytotoxic T lymphocytes in macaques by using a multiepitope gene and DNA prime-modified vaccinia virus Ankara boost vaccination regimen. J Virol. 1999 Sep;73(9):7524-32. doi: 10.1128/JVI.73.9.7524-7532.1999. PMID 10438842